CLINICAL TRIAL: NCT02732405
Title: A Multicenter, Open Label, Pilot Study to Investigate Tolerability and Efficacy of MK5172 / MK8742 Without Ribavirin for 12 Weeks in Patients With Chronic HCV G1b Infection With Compensated Cirrhosis (Child-Pugh A5 to A6) and No Response to PR or Prior Failure to First Generation Protease Inhibitors (PIs)
Brief Title: Study to Investigate Tolerability and Efficacy of MK5172 / MK8742 Without Ribavirin for 12 Weeks in Patients With Chronic HCV G1b Infection With Compensated Cirrhosis
Acronym: GECOM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: CD Pharma Group S.r.l. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004713-24
Record Dates: First submitted 2016-03-15; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C; Compensated Cirrhosis
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK5172 /MK8742 (Experimental)
  Interventions: Drug: MK5172 /MK8742

INTERVENTIONS:
Drug: MK5172 /MK8742 — tablets of MK-5172 100 mg/MK-8742 50 mg will be administered orally, daily for 12 weeks without ribavirin

SUMMARY:
To assess efficacy (SVR rate) of MK5172 / MK8742 for 12 weeks without RBV in G1b patients with compensated cirrhosis (Child-Pugh A5 to A6) previously failing first gen. PI or non responders to PR.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed,
2. Age > 18 years,
3. Chronic infection with Hepatitis C virus genotype 1b,
4. HCV RNA > 100 IU/mL,
5. HCV patients previously treated by PR with no response or previously treated with first generation PIs (boceprevir, telaprevir, simeprevir) and failing therapy,
6. Subjects with compensated cirrhosis with Child-Pugh score ranging between A5 to A6. Cirrhosis defined by liver biopsy (METAVIR F4) or non-invasive methods (transient elastography (FibroScan) > 12.5 KPa; or FibroTest or FibroSure > 0.75 with APRI >2),
7. Hepatic Venous Pressure Gradient (HVPG) > 6 mmHg (only in selected sites),
8. Albumin level ≥ 3.0 g/dl,
9. Platelet count ≥ 75 x 103/μL.

Exclusion Criteria:

1. Child-Pugh score greater than CP-A6,
2. Patients with HCV genotype 1a, 2, 3, 4, 5, 6,
3. Have any serious or active medical illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance,
4. HIV or chronic hepatitis B virus (HBV) infection (HBsAg positive),
5. Decompensated cirrhosis/previous decompensation,
6. Pregnancy,
7. Breast-feeding,
8. Known hypersensitivity to Grazoprevir, Elbasvir or any of its components,
9. Albumin level < 3.0 g/dl,
10. Platelet count < 75 x 103/μl,
11. Concomitant participation in any clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response rates 12 weeks after discontinuation of therapy (SVR12). SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug. | 12 weeks after discontinuation of therapy (SVR12).

IPD SHARING:
Plan to Share IPD: No